CLINICAL TRIAL: NCT02391727
Title: A Phase 1, Multi-center, Open-Label Dose Escalation Study of SYN004 in Patients With Solid Tumors to Evaluate the Safety, Immunogenicity and Pharmacokinetics of SYN004 Following Administration of Eight Intravenous Doses
Brief Title: Safety, Immunogenicity and Pharmacokinetics of SYN004 in Patients With Solid Tumors
Acronym: SYN004_Ph_1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synermore Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYN004-001
Record Dates: First submitted 2015-03-09; First posted 2015-03-18 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Colon Cancer, Breast Cancer, Cancer of the Head and Neck
Keywords: SYN004; cetuximab
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms; Head and Neck Neoplasms | interventions — SYN-004

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SYN004 (Other): open label study
  Interventions: Biological: SYN004

INTERVENTIONS:
Biological: SYN004 — subjects who have received effective treatment for their cancers are eligible

SUMMARY:
A first-in-human evaluation of SYN004, a monoclonal antibody that binds to the EGF receptor on cancer cells. Cetuximab, a marketed antibody, has been shown to be effective by inhibiting the growth of cancer cells thereby prolonging the life of patients who have received it. SYN004 is a closely related monoclonal antibody also binds to the EGF receptor in the same way. SYN004 might also inhibit cancer cells and prolong life but has been engineered to avoid some of the hypersensitivity reactions known to provoked by cetuximab.

DETAILED DESCRIPTION:
Study Design:

In this open-label, dose escalation study, subjects will receive a single IV loading dose of SYN004 on Day 1 of the first treatment week, followed by up to 7 fixed weekly doses of SYN004. Subjects will be assigned to loading and fixed doses by dose group.

Each dose group will comprise 3 subjects and may be expanded to 6 subjects. Subjects will enter dose groups in the order in which they are enrolled. There will be no intra-subject dose adjustments.

Only 1 subject in a cohort may receive the loading dose of SYN004 on any given day; at least 1 day must elapse before the next subject in the cohort receives the loading dose.

Study SYN004-001 Dose Matrix. Three initial subjects will be enrolled followed by an additional three if specified by protocol. Dose levels are specified below.

Group 1: Loading dose: 100 mg/m2; Weekly Dose: 62.5 mg/m2. Group 2: Loading dose: 200 mg/m2; Weekly Dose: 125 mg/m2. Group 3: Loading dose: 400 mg/m2; Weekly Dose: 250 mg/m2.

After each dose of IV SYN004, subjects will be observed in the clinic for 12 hours. After the loading dose, subjects will undergo safety evaluations on Days 2, 3 and 5. Safety evaluation will also be performed on Day 1 (pre-treatment) and Day 3 of each fixed dose treatment week.

Dose-limiting toxicities (DLTs) are defined as any Grade ≥3 AE assessed by the investigator or Medical Monitor, with agreement of the Safety Review Board (SRB), as related to SYN004. Subjects with DLTs will be withdrawn from treatment. If 2 or more subjects in a dose group experience DLTs, or one subject in a dose group experiences a Grade ≥3 infusion reaction, all subjects in that dose group will be withdrawn from treatment.

Subjects in the dose groups are considered evaluable for dose escalation decisions if they receive at least 4 doses of SYN004, or discontinue SYN004 because of a DLT.

Subjects who withdraw or are terminated per protocol before receiving 4 doses of SYN004 will be replaced.

For subjects who receive at least 4 doses of SYN004, End of Study CT scans for RECIST (version 1.1) evaluation will be performed six (6) days following the final SYN004 treatment.

There will be a 28-day safety monitoring period following the final dose of SYN004 for all subjects in the study. All subjects will attend an End-of-Study Visit 28 days after the final dose of SYN004.

Subjects who complete Cycles 1 and 2, who have evidence of improvement per RECIST 1.1 (i.e., findings of complete or partial response per RECIST 1.1) and meet the other eligibility criteria will be offered up to 3 additional treatment cycles (i.e., up to 12 additional weekly doses) of SYN004 in the SYN004-001 Extension Study. During the Extension Study, subjects will receive the same fixed dose of SYN004 they received in Cycles 1 and 2.

Dose escalation will proceed according to a standard 3+3 study design.

ELIGIBILITY:
Inclusion Criteria:

Note: No waivers of the study inclusion or exclusion criteria will be granted.

1. Diagnosis of a solid tumor for which the accepted standard of care includesa licensed anti-EGFR therapy;
2. Tumor progression in patients with RAS wild type metastatic colorectal cancer irrespective of their exposure to licensed anti-EGFR therapy including anti-EGFR antibodies; OR Tumor progression in patients with metastatic colorectal cancer refractory to cetuximab or panitumumab or other anti-EGFR antibodies OR Tumor progression in patients with EGFR-mutated non-small cell lung cancer (NSCLC) who have refused therapy.

   OR Tumor progression or recurrence in patients with squamous cell carcinoma of the head and neck irrespective of their exposure to licensed anti-EGFR therapy including anti-EGFR antibodies.

   OR Patients with locally advanced or metastatic colorectal carcinoma who have
   1. relapsed after standard of care treatment,
   2. proved refractory to standard of care treatment
   3. refused standard of care treatment
   4. been found to be medically unsuitable for standard of care treatment
3. Completion of written informed consent procedure;
4. Male or female subjects over 17 years of age
5. Life expectancy of at least 3 months;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2;
7. At least one measureable non-irradiated site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
8. Adequate bone marrow function, with absolute neutrophil count (ANC) >1,500/mm3, platelet count >100,000/mm3, and hemoglobin > 10 g/mm3;
9. Adequate liver function, with bilirubin <1.5 x the upper limit of the normal range (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x the ULN;
10. Adequate renal function, with serum creatinine <1.5 mg/dL;
11. Adequate cardiac function, with left ventricular ejection fraction (LVEF) ≥50%, normal electrocardiogram, and absence of significant cardiac disease;
12. In women of childbearing potential (defined as women of reproductive capacity who are pre-menopausal or within 12 months of cessation of menses): negative serum pregnancy test and use of an acceptable non-hormonal method of contraception;
13. Ability to communicate with the investigator, and understand and comply with the requirements of the protocol;
14. Agrees to notify the investigator when deviating from the protocol requirements with regard to concomitant medications;
15. Agrees to stay in contact with the study site for the duration of the study and to provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study.

Exclusion Criteria:

1. Participation in a study of an investigational agent or use of an investigational device at the time of screening or within 4 weeks of enrollment;
2. Receipt of treatment with a monoclonal antibody (mAb) within 4 weeks of enrollment or not recovered from an adverse event (i.e., event is >Grade 1 or subject has not returned to baseline) due to treatment with a mAb administered >4 weeks before enrollment;
3. Receipt of chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to enrollment, or not recovered from an adverse event (i.e., event is >Grade 1 or subject has not returned to baseline) due to a previously-administered agent;
4. Major surgical procedure or significant traumatic injury within 4 weeks prior to screening;
5. Diagnosis of an additional malignancy that is progressing and requires treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and in situ cervical cancer that has undergone potentially curative therapy;
6. Active autoimmune disease requiring systemic treatment within the past 3 months, or a documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents (subjects with vitiligo or resolved childhood asthma/atopy are allowed);
7. Diagnosis of an immune deficiency;
8. Receipt of systemic steroids or any form of immunosuppressive therapy within 7 days prior to enrollment, with the following exceptions:

   1. Stable doses of topical, ocular, intranasal or inhaled corticosteroids
   2. Doses of systemic steroids that, in the opinion of the investigator, are pysiologic replacement doses
   3. Systemic steroids as prophylactic treatment for subjects with allergy to contrast media
   4. Non-absorbed intra-articular steroid injections
   5. Systemic corticosteroids required for control of infusion reactions or AEs if doses have been tapered to <10 mg prednisone or equivalent for 2 weeks prior to the first study treatment
9. Evidence of interstitial lung disease or active, non-infectious pneumonitis;
10. Active infection requiring systemic therapy;
11. History of cerebrovascular accident, transient ischemic attack, or subarachnoid hemorrhage within 6 months prior to screening;
12. Active hepatitis B (i.e., hepatitis B surface antigen [HBsAg] positive) or hepatitis C (i.e., hepatitis C virus [HCV] ribonucleic acid [RNA; qualitative] is detected);
13. Serious non-healing wound, ulcer, or bone fracture;
14. Any severe or uncontrolled medical condition or other condition that could affect participation in the study;
15. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 28 days of last SYN004 Administration
  cutaneous toxicity, hypersensitivity

SECONDARY OUTCOMES:
maximum plasma concentration (Cmax) | 84 days
  Cmax will be determined using noncompartmental methods for SYN004
time to Cmax (Tmax) | 84 days
  Tmax will be determined using noncompartmental methods for SYN004
elimination rate constant (λz) | 84 days
  λz will be determined using noncompartmental methods for SYN004
elimination half-life (t½) | 84 days
  t½ will be determined using noncompartmental methods for SYN004
mean residence time (MRT) | 84 days
  MRT will be determined using noncompartmental methods for SYN004
area under the plasma concentration vs. time curve from 0 (initiation of infusion) to the time of the last detectable concentration (AUC0-t), AUC from time 0 extrapolated to infinity (AUC0-∞) | 84 days
  AUC0-t and AUC0-∞ will be determined using noncompartmental methods for SYN004
systemic clearance (CL) | 84 days
  CL will be determined using noncompartmental methods for SYN004
volume of distribution in the terminal phase (Vdβ), and estimated steady-state volume of distribution (VSS) | 84 days
  Vdβ and VSS will be determined using noncompartmental methods for SYN004
anti-cancer activity | 84 days
  Measurement of objective response (OR), durability of objective response (DOR), and progression-free survival (PFS). The number and proportion of subjects who achieve objective tumor response (complete response [CR], partial response [PR], and CR+PR) or stable disease (SD) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, according to local radiological assessments from date of first administration of the investigational product to the end of the study treatment.

OTHER OUTCOMES:
To assess biomarkers of relevance to SYN004 mechanism of action and activity | 84 days
  Blood samples will be collected for the evaluation of IgE antibodies to Galα1,3Gal

CONTACTS AND LOCATIONS:
Overall Officials: John McClain, MD, Study Director — Synermore Biologics Co., Ltd.
Locations (2):
- United States (2):
  - Ochsner Medical Center, New Orleans, Louisiana
  - Washington University Medical Center, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No